CLINICAL TRIAL: NCT05619042
Title: Detection of Coronary Artery Calcifications by Whole Blood Transcriptome Analyzed by Artificial InTelligence Algorithms. (CAC-TRAIT Study)
Brief Title: Detection of Coronary Artery Calcifications by Whole Blood Transcriptome Analyzed by Artificial InTelligence Algorithms
Acronym: CAC-TRAIT
Status: Completed | Type: Observational
Sponsor: Santiago Gabriel Miriuka (Other)
Collaborators: Fundación para la Lucha contra las Enfermedades Neurológicas de la Infancia (Other)
Responsible Party: Sponsor-Investigator, Santiago Gabriel Miriuka, Co-Founder & CEO, MultiplAI Health Limited
Organization: MultiplAI Health Limited (Other)
Other Study IDs: CCT2
Record Dates: First submitted 2022-11-01; First posted 2022-11-16 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Atherosclerosis; Atheroscleroses, Coronary; Atherosclerotic Plaque
Keywords: risk stratification; Cardiovascular disease (CVD) screening; general population; transcriptomics; primary prevention; artificial intelligence; no history of CVD; subclinical
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease; Plaque, Atherosclerotic; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Mouth swab samples, whole blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Presence / absence of CAC: Participants with or without a level/extension of CAC

SUMMARY:
The goal of this observational study is to determine the diagnostic accuracy of peripheral whole blood transcriptomes analyzed by an artificial intelligence algorithm to detect the presence and extent of coronary calcification in individuals without a history of known cardiovascular disease.

The main question it aims to answer is:

1. Will the proposed method predict the presence and extent of coronary artery calcification from the peripheral whole-blood transcriptomes?

DETAILED DESCRIPTION:
This study will be a prospective observational single-site study. A convenience sample will be carried out to include 800 patients who attend the Clinic, to undergo a cardiac CT without contrast (coronary calcium score), either for a medical indication or volunteers for an assessment of cardiovascular risk. The study will have a baseline stage in which a clinical evaluation will be performed, blood samples will be drawn for transcriptome analysis and laboratory analysis. Then, a DNA sample obtained by swabbing the buccal mucosa will be taken. Subsequently, a non-contrast gated cardiac CT will be performed to assess the presence and extent of coronary calcification and other outcomes of interest. At the end of patient enrollment, biological samples will be sequenced for in silico evaluation of the results. Finally, a 5-year clinical (telephone) follow-up will be carried out to collect data on the incidence of fatal and non-fatal cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 30 and 75 years attending the institution for a non-contrast cardiac CT scan (coronary calcium score) either by medical indication or voluntary for cardiovascular risk assessment.
* Signature of the informed consent form

Exclusion Criteria:

* Previously known chronic renal or hepatic insufficiency.
* Active chronic lung disease, defined as exacerbated asthma, exacerbated chronic obstructive pulmonary disease (COPD), or pulmonary fibrosis.
* Active and/or previous cardiovascular disease, defined as previous acute myocardial infarction, stable or unstable angina, cerebrovascular accident, history of vascular interventions (coronary or another territory), heart failure, severe cardiomyopathies, or valvulopathies.
* Uncontrolled hyper or hypothyroidism.
* Suprarenal insufficiency.
* Previous surgeries in the last 3 months.
* Severe trauma in the last 6 months, defined as one that involved bone fractures and/or surgical interventions.
* Known active cancer disease or under treatment (acute or preventive), or history of cancer disease without criteria for a cure.
* Known autoimmune disease active or in treatment.
* Ongoing pregnancy, postpartum period of fewer than 12 months, or breastfeeding.
* Other serious illnesses with an estimated life expectancy of fewer than 12 months (according to the investigators).
* Temperature greater than 37.5°C recorded by a thermometer or any acute infection caused by viruses or bacteria confirmed by a health professional in the previous 30 days.
* Pathologies under immunosuppressive treatment

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women between 30 and 75 years attending the institution for a non-contrast cardiac CT scan (coronary calcium score) either by medical indication or voluntary for cardiovascular risk assessment.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
Coronary artery calcium score | At baseline (cross-sectional assessment)
  Coronary artery calcium (CAC) score (Agatston units) stratified with increasing risk according to the Society of Cardiovascular Computed Tomography Guidelines as CAC=0; CAC 1-99; CAC 100-299; and CAC≥300.

SECONDARY OUTCOMES:
Coronary artery calcium score | At baseline (cross-sectional assessment)
  Percentile Agatston score: according to age and sex with a increasing risk ranging from 1 to 99 th percentile.
Coronary artery calcium score (number of segments) | At baseline (cross-sectional assessment)
  Number of segments with coronary calcifications ranging from 0 to 17 segments.
Aortic valve calcium | At baseline (cross-sectional assessment)
  Aortic valve calcification score (Agatston units) as a continuous variable with increasing risk and without preestablished thresholds
Thoracic aorta calcium | At baseline (cross-sectional assessment)
  Thoracic aorta calcification score (Agatston units) as a continuous variable with increasing risk and without preestablished thresholds
Epicardial adipose tissue (volume) | At baseline (cross-sectional assessment)
  cm2/m2
Epicardial adipose tissue (density) | At baseline (cross-sectional assessment)
  density, Q1-Q4: quartiles percentage
Fatty liver | At baseline (cross-sectional assessment)
  liver attenuation <48 Hounsfield units
Neutrophil to lymphocyte ratio | At baseline (cross-sectional assessment)
  hematological parameter for systemic inflammation and stress
High-sensitive C reactive protein (CRP) | At baseline (cross-sectional assessment)
  mg/dl
Repolarization abnormalities | At baseline (cross-sectional assessment)
  Number of participants with repolarization abnormalities on a 12-lead ECG, defined as ST segment depression or pathological T wave inversion.
Left ventricular hypertrophy | At baseline (cross-sectional assessment)
  Number of participants with left ventricular hypertrophy on a 12-lead ECG, defined by positive Sokolow-Lyon or Cornell criteria.
Intraventricular conduction abnormalities | At baseline (cross-sectional assessment)
  Number of participants with intraventricular conduction abnormalities on a 12-lead ECG, stratified by the presence of left bundle branch
  block; right bundle branch block and left posterior fascicular block; right bundle branch block and left anterior fascicular block or right bundle branch block; or left anterior fascicular block.
Percent electron density relative to water (%EDW) | At baseline (cross-sectional assessment)
  percent electron density relative to water, available for direct evaluation with dedicated software in all scans acquired using a dual-layer spectral CT scanner).
Death | year 1 through 5
  Number of participants with report of death from any cause
Acute ischemic syndrome | year 1 through 5
  Number of participants with non fatal diagnosis of acute myocardial infarction or unstable angina
Heart failure | year 1 through 5
  Number of participants with non fatal new diagnosis of heart failure with preserved or impaired ventricular function
Vascular revascularization | year 1 through 5
  Number of participants with performance of myocardial revascularization surgery, coronary angioplasty or peripheral vascular angioplasty
cerebrovascular event | year 1 through 5
  Number of participants with non fatal diagnosis of cerebrovascular accident ("stroke") or transient ischemic attack
Cancer | year 1 through 5
  Number of participants with new diagnosis of any type of cancer

CONTACTS AND LOCATIONS:
Overall Officials: Santiago G Miriuka, MD MSc PhD, Principal Investigator — MultiplAI Health LTD
Locations (1):
- Clinica Sagrada Familia, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-12): https://cdn.clinicaltrials.gov/large-docs/42/NCT05619042/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-06): https://cdn.clinicaltrials.gov/large-docs/42/NCT05619042/ICF_001.pdf